CLINICAL TRIAL: NCT01090349
Title: CLINICAL EVALUATION OF REMOTE MONITORING WITH DIRECT ALERTS TO REDUCE TIME FROM EVENT TO CLINICAL DECISION. (REACT Study)
Brief Title: Clinical Evaluation Of Remote Monitoring With Direct Alerts To Reduce Time From Event To Clinical Decision
Acronym: REACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CR-09-064-WW-RC
Record Dates: First submitted 2010-03-18; First posted 2010-03-19 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: The Patient Meets ACC/AHA/ESC Guidelines for Implantable Cardioverter Defibrillator (ICD) or Cardiac Resynchronization Therapy (CRT-D) Device
Keywords: ICD, CRTD, Remote Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Direct Alerts ON (Experimental): Direct Alerts in implantable device were turned on
  Interventions: Device: Implantation of an ICD/CRT-D device; Device: Merlin.NET PCN
- Direct Alerts OFF (Active Comparator): Direct Alerts in implantable device were turned off
  Interventions: Device: Implantation of an ICD/CRT-D device; Device: Merlin.NET PCN

INTERVENTIONS:
Device: Implantation of an ICD/CRT-D device — The Implantable Cardioverter Defibrillator (ICD) or Cardiac Resynchronization Therapy (CRT-D) device and leads are not the devices being evaluated in this investigation.
  Other Names: The SJM ICD family of devices with the Invisilink feature are the AnalyST™ and /AnalyST Accel™ and Current™/CurrentTM RF/Current AccelTM.; The SJM CRT-D family of devices with the Invisilink feature is the Promote™/PromoteTM RF.
Device: Merlin.NET PCN — The Merlin.Net™ PCN is a dedicated computer system that connects physicians to patients outside of the clinic setting by centralizing data from remote transmissions, implant procedures and in-clinic follow-ups into single location with easy export to Electronic Health Record (EHR) systems
  Other Names: Merlin.NET

SUMMARY:
St. Jude Medical developed the Merlin.net™ Patient Care Network (Merlin.net™ PCN) to augment or replace routine scheduled in-clinic visits.

This investigation is designed with the hypothesis that detection of events (system integrity and diagnostic related) through Direct Alerts™ via Remote Monitoring allow clinicians an earlier opportunity to address and resolve events and may therefore improve patient care.

ELIGIBILITY:
Inclusion Criteria:

* The patient meets ACC/AHA/ESC guidelines for implantable cardioverter defibrillator (ICD) or cardiac resynchronization therapy (CRT-D) device
* The patient is recently (≤2 weeks) implanted with a SJM device compatible with the Merlin.net™ PCN - (inclusive of upgrade from ICD to CRT-D or an implantable pulse generator change)
* The patient has a life expectancy of greater than 12 months (based on the physician's discretion).
* The patient is mentally capable to participate in the investigation (based on the physician's discretion).
* The patient is 18 years of age or older

Exclusion Criteria:

* The patient is being actively considered for cardiac transplantation.
* The patient has primary valvular disease that has not been corrected.
* The patient had a myocardial infarction within the last month
* The patient had unstable angina within the last month.
* The patient has had Coronary Artery Bypass Grafting (CABG) within the last month.
* The patient had a Percutaneous Coronary Angioplasty (PTCA) within the last month.
* The patient is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2010-03; Primary Completion 2012-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
time between the detection of an event and the point in time when the physician or delegate takes a clinical decision | 2 years

SECONDARY OUTCOMES:
The sufficiency of the device data retrieved through the Remote Monitoring feature to make a clinical decision | 2 years
The physician or delegate time required for remote follow up as compared to in-clinic follow up | 2 years
The changes over one year in the Hospital Anxiety and Depression Scale (HADS) for the two different randomization arms | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Janet McComb, MD, Principal Investigator — Freeman Hospital Newcastle; UK
Locations (2):
- Dr. Ralph Bosch, Ludwigsburg, Germany
- Freeman Hospital, Newcastle, United Kingdom